CLINICAL TRIAL: NCT02752607
Title: The STEP-CAT Cohort Management Study: Step-down to Prophylactic Doses of Enoxaparin After a Minimum of 3-6 Months of Anticoagulation for the Treatment of Cancer-associated Thrombosis.
Brief Title: Reduction to Preventive Doses of Enoxaparin After 3 to 6 Months of Treatment With Blood Thinners for Cancer-associated Blood Clots
Acronym: STEP-CAT
Status: Terminated | Type: Observational
Why Stopped: The study was stopped early due to low recruitment
Sponsor: Dr. Vicky Tagalakis (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Dr. Vicky Tagalakis, Attending Physician and Clinical Researcher, Lady Davis Institute
Organization: Lady Davis Institute (Other)
Other Study IDs: MM-JGH-16-003
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background: Venous thromboembolism (VTE), which includes deep vein thrombosis (DVT) and pulmonary embolism (PE), is the third most common cardiovascular disorder after myocardial infarction and stroke. VTE occurs in about 1 person per 1,000 per year, increasing dramatically in patients with cancer to about 25 per 1,000 per year. Among the known risk factors of VTE, cancer is one of the most potent. Patients with cancer have a 7- to 28-fold higher risk for VTE than non-cancer patients. VTE has important implications for the care of cancer patients, including reduced life expectancy, high rates of VTE recurrence both while on and after stopping anticoagulation, the need for chronic anticoagulation with related adverse drug reactions, and delays in cancer therapies. Clinical dilemma: Current clinical guidelines recommend a minimum of 3-6 months of anticoagulation with weight-adjusted low molecular weight heparin (LMWH) in cancer patients with VTE. However, there are no recommendations beyond the initial 6 months of therapy due to the lack of data on extended duration therapy for cancer-associated thrombosis (CAT). This leads to variability in physician practices, with some continuing weight-adjusted LMWH therapy beyond 6 months. This poses concern because, while the goal is to prevent recurrence of VTE, the risk of major bleeding with prolonged weight-adjusted LMWH therapy is significant. Potential solutions: There is a lack of data to inform on VTE treatment in cancer patients beyond the initial 3-6 months of anticoagulation. We propose that after a minimum of 3-6 months of therapeutic dose anticoagulation, the use of prophylactic doses of LMWH will have an acceptable and adherence profile in cancer patients with VTE. The data obtained from this study will help inform physician practices. Design: This is a multicentre, open-label study of enoxaparin (40 mg subcutaneous injection, once daily) for additional 6 months after an initial minimum 3-6-month course of therapeutic dose anticoagulant therapy. Patients: 150 patients with VTE secondary to cancer will take part in this multicentre study conducted in 8 Canadian centres within Quebec, Ontario and Nova Scotia. Study Outcomes: The primary objective of the study is to determine the rate of recurrent VTE in patients receiving prophylactic dose enoxaparin for secondary VTE prophylaxis after an initial minimum 3-6 months of anticoagulation. The secondary objective is to determine the safety profile of prophylaxis dose enoxaparin for secondary VTE prophylaxis after an initial 3-6 months of anticoagulation. This includes determining for all subjects: 1) cumulative incidence of major bleeding events; 2) cumulative incidence of clinically relevant non-major bleeding events; 3) cumulative incidence of minor bleeding event, and 4) overall survival during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have an active malignancy defined as any of: a) Diagnosis of cancer (excluding basal cell or squamous cell carcinoma of the skin) within 18 months of enrollment; b) Have received treatment for cancer within 18 months (e.g. radiation therapy, chemotherapy, adjuvant therapy); c) Have documented recurrent or metastatic cancer
* Receiving a 3-6 month course of weight-adjusted LMWH for an acute, objectively confirmed, symptomatic VTE (proximal or distal DVT of the lower extremity, proximal DVT of the upper extremity, or PE)
* Age ≥ 18 years
* Life expectancy > 6 months
* Able to comply with scheduled follow up visits
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Willing to provide written informed consent

Exclusion Criteria:

* Distal DVT of the upper extremity
* Recurrent VTE during the 3-6-month LMWH treatment period
* Major or clinically relevant non-major bleeding during the 3-6 month LMWH treatment period
* Risk of bleeding (e.g. recent neurosurgery, history of intracranial hemorrhage, acute gastroduodenal ulcer, etc.)
* Diagnosis of basal cell and squamous cell carcinoma of the skin or acute Leukemia
* Platelet count < 50 x 109/L
* Creatinine clearance <30ml/min (using the modified Cockcroft-Gault formula)
* On hemodialysis
* Known hypersensitivity to heparin, LMWHs, or pork products
* Known contraindication to the use of heparin (e.g. heparin-induced thrombocytopenia)
* Currently participating in another clinical trial involving anticoagulation therapy (with the exception of aspirin)
* Pregnancy or breastfeeding
* On an anticoagulant for a different indication
* Treating physician plans for weight-adjusted LMWH for longer than 3-6 months duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will have an active malignancy defined as any of: a) diagnosis of cancer (excluding basal cell or squamous cell carcinoma) within 18 months of study enrolment; or b) have received treatment for cancer within 18 months (e.g. radiation therapy, chemotherapy, adjuvant therapy) of study enrolment; or c) have documented recurrent or metastatic cancer. Subjects must also have a first episode of objectively confirmed VTE (distal or proximal deep vein thrombosis (DVT) of the lower limb or proximal DVT of the upper limb, or pulmonary embolism (PE)) that is being treated with therapeutic anticoagulation for a minimum intended duration of 3-6 months. Subjects must be ≥18 years of age with a life expectancy of > 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-05; Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Rate of recurrent VTE | 6 months

SECONDARY OUTCOMES:
Cumulative incidence of major bleeding events | 6 months
Cumulative incidence of clinically relevant non-major bleeding events | 6 months
Cumulative incidence of minor bleeding events | 6 months
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Tagalakis, MD, MSc, Study Chair — The Lady Davis Insitute, Jewish General Hospital
Locations (7):
- Canada (7):
  - Queen Elizabeth II Medical Centre, Halifax, Nova Scotia
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Hôpital Charles-Le Moyne, Greenfield Park, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - St-Mary's Hospital, Montreal, Quebec
  - The McGill University Health Centre - Glen Site, Montreal, Quebec
  - Hôpital Sacré-Coeur, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Popov J, Coelho S, Carrier M, Sperlich C, Solymoss S, Routhier N, Shivakumar S, Aibibula W, Kahn SR, Tagalakis V. Step down to 6 months of prophylactic-dose low molecular weight heparin after initial full-dose anticoagulation for the treatment of cancer-associated thrombosis (STEP-CAT): A pilot study. J Thromb Haemost. 2022 Aug;20(8):1868-1874. doi: 10.1111/jth.15760. Epub 2022 Jun 9. PMID 35587536